CLINICAL TRIAL: NCT04074577
Title: Computer Aided Detection, Tandem Colonoscopy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-00801
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Technique followed by Combination (Active Comparator): Back-to-back tandem colonoscopies by the same endoscopist using an Olympus 190 colonoscope. The first colonoscopy will be performed without automated polyp detection software (standard technique) followed immediately by another colonoscopy with automated polyp detection software (combination technique).
  Interventions: Diagnostic Test: Standard technique First
- Combination +followed by Standard Technique (Active Comparator): Back-to-back tandem colonoscopies by the same endoscopist using an Olympus 190 colonoscope. In this arm, the first colonoscopy with be performed with automated polyp detection software (combination technique) followed immediately by another colonoscopy without automated polyp detection software (standard technique)
  Interventions: Diagnostic Test: combination technique First

INTERVENTIONS:
Diagnostic Test: Standard technique First — colonoscopy without automated polyp detection software
  Arms: Standard Technique followed by Combination
Diagnostic Test: combination technique First — automated polyp detection software
  Arms: Combination +followed by Standard Technique

SUMMARY:
The purpose of this project is to examine the role of machine learning and computer aided diagnostics in automatic polyp detection and to determine in real-time how a computer-aided detection (CADe) algorithm will perform when compared to standard screening or surveillance colonoscopy alone. Design will be a multi-center, prospective, unblinded randomized tandem colonoscopy study. 196 patients referred for either screening or surveillance colonoscopy will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the endoscopy unit for a screening colonoscopy or a surveillance colonoscopy
* Willingness to undergo tandem colonscopies with and without the use of computer-aided software while undergoing conventional colonoscopy with sedation
* Ability to provide written, informed consent (approved by IRB) and understand the responsibilities of trial participation

Exclusion Criteria:

* People with diminished cognitive capacity
* Patients undergoing diagnostic colonoscopy (e.g. as an evaluation for active GI bleed)
* Patients with incomplete colonoscopies (those where endoscopists did not successfully intubate the cecum due to technical difficulties or poor bowel preparation)
* Patients that have standard contraindications to colonoscopy in general (e.g. documented acute diverticulitis, fulminant colitis and known or suspected perforation).
* Patients with inflammatory bowel disease
* Patients referred for endoscopic mucosal resection (EMR)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Number of adenomas detected in combination technique compared to adenomas detected in standard technique Measured by Adenoma Miss Rate (AMR) | 1 Year
  AMR will be calculated as the number of adenomas detected on the second pass or portion in either group divided by the total number of adenomas detected during both passes.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Gross, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States